CLINICAL TRIAL: NCT07357974
Title: Impact of Sotatercept on Pulmonary Artery and Right Ventricle Remodeling Imaging Assessed With 68Ga-FAPI PET/CT in Patients With PAH: a Pilot Study
Brief Title: Impact of Sotatercept on Pulmonary Artery and Right Ventricle Remodeling Imaging Assessed With 68Ga-FAPI PET/CT in Patients With PAH
Acronym: SOFAPI
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC24.0296
Record Dates: First submitted 2025-12-02; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: [68Ga]Ga-FAPI PET/CT (FAPI); [68Ga]Ga-MAA lung perfusion PET/CT
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: This pilot study explores innovative imaging techniques, including [⁶⁸Ga]Ga-FAPI PET/CT and [⁶⁸Ga]Ga-MAA lung perfusion PET/CT , which have not yet been fully evaluated in patients with pulmonary arterial hypertension.
  Patients with an indication for sotatercept will be screened for eligibility according to predefined inclusion criteria. Eligible participants will be enrolled in the study. Each participant will undergo a comprehensive assessment including [⁶⁸Ga]Ga-FAPI PET/CT and [⁶⁸Ga]Ga-MAA PET/CT at baseline and at a follow-up visit 24 weeks later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/CT (Experimental)
  Interventions: Diagnostic Test: [68Ga]Ga-FAPI PET/CT; Diagnostic Test: [68Ga]Ga-MAA PET/CT

INTERVENTIONS:
Diagnostic Test: [68Ga]Ga-FAPI PET/CT — [68Ga]Ga-FAPI PET/CT
Diagnostic Test: [68Ga]Ga-MAA PET/CT — [68Ga]Ga-MAA PET/CT

SUMMARY:
Pulmonary arterial hypertension (PAH) is a rare, progressive disease characterized by structural changes in the pulmonary arteries, leading to increased pulmonary vascular resistance and elevated pulmonary arterial pressure and, if untreated, right heart failure. Diagnosis requires a comprehensive evaluation, including right heart catheterization performed in specialized centers.

Despite advances in the understanding and management of the disease, PAH remains a severe condition. Current approved therapies primarily target three key pathways involved in endothelial dysfunction: the endothelin, nitric oxide, and prostacyclin pathways. Pulmonary arterial remodeling is characterized by alterations in endothelial cells, smooth muscle cells, and fibroblasts, with fibroblast activation and macrophage involvement contributing to disease progression.

Two positron emission tomography/computed tomography (PET/CT) imaging approaches are currently under investigation in PAH. [⁶⁸Ga]Ga-FAPI PET/CT targets activated fibroblasts and enables noninvasive assessment of fibroblast activity and tissue remodeling. [⁶⁸Ga]Ga-MAA lung perfusion PET/CT is an emerging imaging technique that provides higher spatial resolution and sensitivity than conventional lung perfusion imaging and allows evaluation of regional pulmonary perfusion.

Sotatercept is a novel fusion protein that modulates signaling within the transforming growth factor-beta (TGF-β) superfamily by binding select ligands involved in vascular remodeling. Its mechanism of action is distinct from that of currently approved PAH therapies. Sotatercept has been evaluated in clinical development programs, including the PULSAR and STELLAR studies. Reported adverse events include epistaxis, dizziness, increased hemoglobin levels, and changes in blood pressure.

This study is designed with the following objectives:

Primary objective: To assess pulmonary vascular remodeling in patients with PAH using [⁶⁸Ga]Ga-FAPI PET/CT imaging.

Secondary objectives: To evaluate [⁶⁸Ga]Ga-FAPI uptake and regional lung perfusion using [⁶⁸Ga]Ga-MAA lung perfusion PET/CT imaging at predefined study time points.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Documented diagnostic right heart catheterization (RHC) within 12 months of screening documenting a minimum PVR of ≥ 4 Wood units and pulmonary capillary wedge pressure (PCWP) or left ventricular end-diastolic pressure (LVEDP) of ≤ 15 mmHg, with the diagnosis of WHO PAH Group 1 in any of the following subtypes:

  * Idiopathic PAH
  * Heritable PAH
  * Drug/toxine-induced PAH
  * PAH associated with connective tissue disease
  * PAH associated with simple, congenital systemic-to- pulmonary shunts at least 1year following repair
* Patients under bi or tri-background-therapy
* Symptomatic PAH classified WHO FC II or III
* Patients will be started on Sotatercept
* Ability to adhere to study visit schedule and understand and comply with all the protocol requirement.
* Ability to understand and provide written informed consent

Exclusion Criteria:

* Diagnosis of PH WHO Groups 2, 3, 4, or 5
* Diagnosis of the following PAH Group 1 subtypes: human immunodeficiency virus (HIV)-associated PAH, PAH associated with portal hypertension, schistosomiasis associated PAH, pulmonary veno occlusive disease and pulmonary capillary hemangiomatosis.
* Hemoglobin at screening above gender-specific ULN, per local laboratory test
* Pregnant or breastfeeding women
* Any of the following clinical laboratory values at the Screening visit:

  * eGFR < 30 mL/min/1.73 m2 (as defined by MDRD equation)
  * Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin levels > 3 × ULN
  * Platelet count < 50,000/mm3 (< 50.0 × 109/L)
* Known allergic reaction to sotatercept (ACE-011), its excipients, or luspatercept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Vascular remodeling as assessed by [68Ga] Ga-FAPI uptake of pulmonary arteries on PET/CT imaging. | at baseline
  A positive uptake will be defined as a ratio of the Standardized uptake value (SUV) max of the pulmonary arteries and the SUVmean of the vascular background activity measured at the center of the left ventricle greater than 1.5.

SECONDARY OUTCOMES:
Change from baseline in [68Ga] Ga-FAPI uptake on pulmonary arteries as assessed by SUVmax at 24 weeks. | At baseline and at 24 weeks.
  [68Ga] Ga-FAPI uptake on pulmonary arteries. This will be assessed using a visual scale and the Standardized uptake value (SUVmax).
Visual assessment of pulmonary artery [68Ga]Ga-FAPI uptake | At baseline and at 24 weeks.
  Change from baseline in regional lung perfusion as assessed by the Pulmonary vascular obstruction index (PVOI) (in %) on [68Ga]Ga-MAA lung perfusion PET/CT imaging at 24 weeks.
[68Ga] Ga-FAPI uptake on the right ventricule (RV) assessed by SUVmax at 24 weeks. | At week 24
RV ventricule dysfunction based on Tricuspid annular plane systolic excursion (TAPSE)<17mm at 24 weeks. | At 24 weeks.
Change from baseline in [68Ga] Ga-FAPI uptake on the RV as assessed by SUVmax at 24 weeks. | At baseline and at 24 weeks.
Mean pulmonary arterial pressure (mPAP) (in mmHg) at baseline. | At baseline.
  mPAP will be measured by right Heart catheterism (RHC).
Cardiac output (CO) (l/mn) at baseline. | At baseline.
  CO will be measured by RHC.
Right atrial pressure (RAP) (mmHg) at baseline. | at baseline
  RAP will be measured by RHC.
Right ventricular pressure (RVP) (mmHg) at baseline. | At baseline.
  CO will be measured by RHC.
Pulmonary vascular resistance (PVR) (Wood unit) at baseline. | At baseline.
  CO will be measured by RHC.
Mean pulmonary arterial pressure (mPAP) (mmHg) at 24 weeks. | At 24 weeks.
  mPAP will be measured by right Heart catheterism (RHC).
Cardiac output (CO) (l/mn) at 24 weeks. | At 24 weeks.
  CO will be measured by RHC.
Right atrial pressure (RAP) (mmHg) at 24 weeks. | At 24 weeks.
  RAP will be measured by RHC.
Right ventricular pressure (RVP) (mmHg) at 24 weeks. | at baseline
  CO will be measured by RHC.
6 minutes walking test result (6MWT) (meters) at baseline. | At baseline.
Vascular remodeling on [68Ga]Ga-FAPI PET/CT is correlated with Nt-proBNP measure in PAH patients | at baseline
  [68Ga] Ga-FAPI uptake on pulmonary arteries (SUVmax) will be correlated with Nt-proBNP measure in PAH patients
6 minutes walking test result (6MWT) (meters) at 24 weeks. | At 24 weeks.
NYHA functional class at baseline. | At baseline.
  The New York heart association (NYHA) scale will be used to classify the severity of the heart failure impact. Classes are defined as I, II, III, IV, with IV indicating severe limitations
NYHA functional class at 24 weeks. | At 24 weeks.
  The New York heart association (NYHA) scale will be used to classify the severity of the heart failure impact extent of heart failure. Classes are defined as I, II, III, IV, with IV indicating severe limitations.
N-terminal pro B natriuretic peptide (NT-pro-BNP) (pg/ml) at baseline | At baseline.
  biological mark indicating heart failure and impact on PH prognosis
N-terminal pro B natriuretic peptide (NT-pro-BNP) (pg/ml) at 24 weeks. | At 24 weeks.
  biological mark indicating heart failure and impact on PH prognosis
Quality of life (QOL) assessed by emPHasis-10 scale at baseline. | At baseline.
  The emPHasis-10 ranges from 0 to 50, with a higher score indicating a poorer health status and QOL.
QOL assessed by emPHasis-10 scale at 24 weeks. | At 24 weeks.
  The emPHasis-10 ranges from 0 to 50, with a higher score indicating a poorer health status and QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Tromeur, Principal Investigator — CHU BREST
Locations (1):
- Chu Brest, Brest, Finistere, France